CLINICAL TRIAL: NCT01262157
Title: A Clinical Randomized Double Blind Placebo Controlled Study on the Effect of Low Intensity Shock Wave Therapy for Erectile Dysfunction in a Group of Patients Not Responding to Oral Therapy
Brief Title: Low Intensity ShockWave Therapy for ED in Non Responders to PDE5i - a Double Blind Placebo Controlled Study
Acronym: LI-ESWT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Yoram Vardi, Rambam Health Care Campus
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 507-10 RMB
Record Dates: First submitted 2010-07-11; First posted 2010-12-17 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; PDE5 Inhibitor; Low intensity shock wave therapy.
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Sham Comparator): We use the same probe that induces the same sensation on the penis and the same noise yet no energy
  Interventions: Device: Extracorporeal Shockwave Therapy Generator (Vascuspec)
- Shock wave therapy (Active Comparator): 12 treatment sessions twice a week during 9 weeks with an interim of 3 weeks no treatment
  Interventions: Device: Low intensity shock wave therapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy Generator (Vascuspec) — Gel is spread around the penis and on the Shock Wave applicator and Treatment (12 sessions in total) of 300 shocks per site, on 5 penile anatomical sites.
  Other Names: Low intensity shock wave Therapy; Extracorporeal Shockwave Therapy
  Arms: placebo
Device: Low intensity shock wave therapy — Gel is spread around the penis and on the Shock Wave applicator and Treatment (12 sessions in total) of 300 shocks per site, on 5 penile anatomical sites.
  Other Names: Low Intensity Extra Corporal Shock Wave Therapy
  Arms: Shock wave therapy

SUMMARY:
Low intensity shock waves (LISW) have been proven in animal studies to induce local growth of new blood vessels. The investigators hypothesized that LISW therapy could improve the symptoms of patients with erectile dysfunction resulting from a problem of blood supply that do not respond to oral therapy (PDE-5 inhibitors).

DETAILED DESCRIPTION:
In this study Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered directly to the penile tissue using a specially designed shockwave device and probe. Shock wave therapy is applied twice a week for three weeks , then a 3- week interval with no therapy followed by another 3 week period of twice a week shock wave therapy. Before and after sexual function questionnaires and objective measures of erectile function will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ED of more than 6 months
* Rigidity score < 3 during PDE5i therapy
* SHIM <21 during PDE5i therapy
* Non- hormonal, neurological or psychological pathology Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Prior prostatectomy surgery
* Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Radiotherapy in pelvic region

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-ED Domain | 17 weeks
  A change of 5 points or more will indicate success

SECONDARY OUTCOMES:
rigidity score | 17 weeks
  a scale of 3 and above indicates success

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Vardi, prof, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel, Israel